CLINICAL TRIAL: NCT01356758
Title: Cardiovascular Risk Assessment in Patients With Severe Psoriasis Treated With Biologic Agents
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Aage Bangs Fond (Other); AbbVie (Industry); Region Midt Forskningsfond (Unknown)
Responsible Party: Sponsor
Other Study IDs: j-nr 20100249
Record Dates: First submitted 2011-05-09; First posted 2011-05-19 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2014-08

CONDITIONS: Psoriasis; Atopic Dermatitis; Atherosclerosis
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic; Atherosclerosis | interventions — Adalimumab; Etanercept; Infliximab; Ustekinumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and skin samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Psoriasis topical treatment: Psoriasis topical treatment. No systemic drugs.
- Psoriasis biological treatment: Psoriasis biological treatment. Anti-Tnf and anti-il12/23.
  Interventions: Drug: biological treatment
- Severe atopic dermatitis: Severe atopic dermatitis
- Control: No intervention. No inflammatory skin disease.

INTERVENTIONS:
Drug: biological treatment — patients treated with anti-psoriatic biological agents
  Other Names: Adalimumab; Etanercept; Infliximab; Ustekinumab
  Groups: Psoriasis biological treatment

SUMMARY:
Psoriasis is a common inflammatory disease of the skin and joints with a prevalence of 1-3% in the caucasian population of Northern Europe and the US. Similarly to other inflammatory diseases there is now substantial and accumulating evidence that psoriasis has a systemic inflammatory component.

It is known that patients suffering from psoriasis have increased prevalence of traditional cardiovascular risk factors, such as hypertension, dyslipidaemia, obesity, tobacco use and diabetes mellitus. This would logically explain an increased rate of cardiovascular events, but even when adjusting for theses risk factors, psoriasis carry an independent risk for developing cardiovascular disease.

Recent large epidemiological studies have shown a strong correlation between psoriasis and myocardial infarction.

Atopic dermatitis has been linked to ischemic stroke in one study, but besides this, the disease has not been associated with cardiovascular disease.

In conclusion, convincing and increasing evidence is supporting that psoriasis induce accelerated atherosclerosis and hence cardiovascular disease and mortality. In particular, this is seen in young patients with early disease onset.

Psoriasis is believed to be driven by cytokines produced by Th1 and Th17 lymphocytes. A number of these cytokines are suggested to be atherogenic. In contrast, another chronic inflammatory disease, atopic dermatitis, is predominantly driven by Th2 lymphocyte derived cytokines, some of which may inhibit atherosclerotic processes. It is therefore, of interest to compare the presence of cardiovascular disease in these two inflammatory skin diseases.

Hypothesis: That the risk of developing cardiovascular disease and especially coronary artery disease is increased in psoriasis patients and that this process can be influenced by treatment of psoriasis with biological treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 years or above.
2. Intervention group: Severe plaque psoriasis with indication for biological therapy according to national guidelines. Psoriasis Control group: Patients with similar disease activity who for personal reasons decline systemic treatment and only receive topical therapy. Atopic dermatitis group: Patients matched regarding sex, disease duration, body surface involvement, BMI and smoking habits.
3. Signed informed consent form prior to initiation of any study-mandated procedure.

Exclusion Criteria:

1. Significant arterial hypertension, unless well controlled with anti-hypertensive medication for at least 1 month before inclusion.
2. Lipid-lowering treatment, unless well controlled for at least 1 month before inclusion.
3. Congestive heart failure (NYHA group III and IV).
4. Reduced kidney function (eGFR below 60).
5. Oral methotrexate, ciclosporin, acitretin and fumarate esters within 1 month before inclusion. In the intervention group, patients receiving oral anti-psoriatic treatment for at least 6 months before the study start can be included, if they are maintained on the same dose during the study period.
6. UVB phototherapy and PUVA photochemotherapy within 1 month prior to study start.
7. Prior treatment with infliximab, etanercept, adalimumab or ustekinumab unless less than PASI-50% reduction have been observed during this treatment.
8. Investigational biological agents within 6 months prior to inclusion.
9. Any other investigational drug within 1 month or 5 half lives prior to inclusion, which ever is longer.
10. Concurrent immunosuppressive or anti-inflammatory treatment for immune diseases other than psoriasis and psoriatic arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with severe psoriasis recruited from a dermatological in- and out patient clinic. Patients with severe atopic dermatitis.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2011-03; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in coronary calcium score (CAC score) | baseline: 0 months, and follow-up: approximately 12 months
  Psoriasis groups evaluated at 0 and approximately 12 months. AD group and controls at baseline only.
Repeated Coronary CT Angiography (CCTA) | 0 and approximately 12 months
  Assessment according to the 18-segment model (as suggested by AHA): Changes in number of coronary plaques, stenosis, severity, composition. Changes in coronary plaque volume index.
  Psoriasis groups evaluated at 0 and approximately 12 months. AD group and untreated controls at baseline only.

SECONDARY OUTCOMES:
Cardiovascular risk markers | 0, 3 and 12 months
  hs-crp, homocystein, SBHG, apolipoprotein B, MBL, PAPP-A.
interleukines in blood | 0, 3 and 12 months
  selected cytokines (amongst: TNFα, IL-1, IL-6, IL-8, IL-10, IL-12, IL-13, IL-15, IL17A, IL-19, IL-20, IL-23, IFN, ICAM-1, E-selectin)
traditional cardiovascular risk factors | 0, 3 and 12 months
  monitoring of blood cholesterol levels and blood glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Kasper F Hjuler, M.D., Principal Investigator — Aarhus University Hospital
Locations (1):
- Dep. of Dermatology, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hjuler KF, Bottcher M, Vestergaard C, Deleuran M, Raaby L, Botker HE, Iversen L, Kragballe K. Increased Prevalence of Coronary Artery Disease in Severe Psoriasis and Severe Atopic Dermatitis. Am J Med. 2015 Dec;128(12):1325-34.e2. doi: 10.1016/j.amjmed.2015.05.041. Epub 2015 Jun 18. PMID 26093174